CLINICAL TRIAL: NCT03205397
Title: Impact of a Child-Parent Preoperative Accompanying Procedure on the Anxiety of Children Aged 5 to 12 With Scheduled Surgery
Acronym: I-PPOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: I15004
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2018-02

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accompanying and information procedure (Experimental): Preparation for anesthesia (explanations, film, booklet), the presence of a relative in the operating room and the awakening of the child.
  Interventions: Other: Experimental Group
- Usual care (Other): Consultation of anesthesia and the care of the child without parental presence
  Interventions: Other: usual care

INTERVENTIONS:
Other: Experimental Group — Preparation for anesthesia (explanations, film, booklet), the presence of a parent in the operating room and the awakening of the child
  Arms: Accompanying and information procedure
Other: usual care — Usual care
  Arms: Usual care

SUMMARY:
In France, during surgery, only 4% of parents are present at induction, most often for children with disabilities with iterative interventions. Some studies have shown that the presence of parents during induction decreases the anxiety of children, while others do not. Their conclusions all advocate preparing parents for this presence in the operating room in an accompanying course.

ELIGIBILITY:
Inclusion Criteria:

* 5 to 12 year olds requiring scheduled surgery
* scheduled outpatient or weekly hospitalization.
* Anesthesia envisaged by inhalation induction
* Agreement of parents (and child according to age).
* Even parent (s) present at pre-anesthesia and on the day of surgery

Exclusion Criteria:

* Child with previous surgery
* Parent (s) of a child who has already had surgery
* Parent (s) or child unable to follow the whole procedure (autism, blindness ...)

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Level of anxiety | 10 minutes
  Level of anxiety measured at the time of anesthetic induction by the MYPAS hetero-evaluation scale

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results of the research — https://www.unilim.fr/reasci/194